CLINICAL TRIAL: NCT04862468
Title: Perivenous Dexamethasone Therapy: Examining Reduction of Inflammation After Thrombus Removal to Yield Benefit in Acute Femoropopliteal DVT (DEXTERITY-AFP)
Brief Title: Perivenous Dexamethasone Therapy: Examining Reduction of Inflammation After Thrombus Removal to Yield Benefit in Acute Femoropopliteal DVT
Acronym: DEXTERITY-AFP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mercator MedSystems, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIP0217; R44HL160434 (NIH)
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Thrombosis, Deep Vein; Iliofemoral; Thrombosis
MeSH Terms: conditions — Venous Thrombosis; Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Combination Product: Perivascular dexamethasone
- Control (Sham Comparator)
  Interventions: Combination Product: Perivascular sham

INTERVENTIONS:
Combination Product: Perivascular dexamethasone — Dexamethasone delivery around target vein segment(s)
  Arms: Treatment
Combination Product: Perivascular sham — Saline delivery around target vein segment(s)
  Arms: Control

SUMMARY:
This is a study of a medical procedure that utilizes a commercially available catheter (the Bullfrog® Micro-Infusion Device) to locally deliver a commercially available anti-inflammatory drug (dexamethasone sodium phosphate injection) around the deep veins after DVT recanalization, where DVT symptoms were present for up to 14 days prior to recanalization. The goal of the study is to see if local anti-inflammation helps prevent re-thrombosis of the blood vessel and improvement in symptoms for up to 24 months after the initial DVT recanalization procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form prior to receiving any non-standard of care, protocol-specific procedures.
2. Stated willingness to comply with all study procedures including completion of questionnaires and follow-up visits and availability for the duration of the study.
3. Male or female, aged 18 to 89 years.
4. For females of reproductive potential: use of highly effective contraception (abstinence is acceptable) for at least 1 month prior to study treatment (unless they had given birth within the 1 month prior to study treatment), and agreement to use such a method for at least 30 days after study treatment.
5. Onset of acute DVT symptoms of 14 days or less prior to initial intervention in the study limb.
6. Ability to take oral medication and be willing to adhere to the prescribed anti-coagulant regimen.
7. Post-procedural prescription for at least 28 days low molecular weight heparin followed by therapeutic anticoagulant of investigator's choice for 12 months minimum as part of post-interventional medication regimen.
8. Minimum of 28 days of prescribed antiplatelet agent (aspirin or P2Y12 inhibitor) for patients receiving stents.
9. DVT located in any of the major femoropopliteal veins (common femoral, femoral, and/or popliteal above the tibial plateau), with possible extension downstream into the iliac veins.
10. Successful recanalization of the target vein with removal of acute thrombus.

Exclusion Criteria:

1. Current enrollment in another non-registry clinical study of systemic drug therapy or another device study that has not completed its primary endpoint, including prior enrollment in this study. Concurrent enrollment in registry studies of approved devices or drugs are acceptable.
2. Lack of capability of understanding the nature, significance and implications of the clinical trial.
3. Body Mass Index between 40 kg/m2 and 45 kg/m2, with significant comorbidity which, in the Investigator's discretion, could impair follow-up or study outcomes.
4. Body Mass Index > 45 kg/m2.
5. Non-ambulatory status prior to DVT occurrence.
6. In the study leg: current established PTS (Villalta ≥ 5 for more than 14 days), current known symptomatic deep venous insufficiency for more than 14 days, or previous symptomatic DVT within the last 365 days.
7. In the contralateral (non-study) leg: symptomatic DVT that, in the opinion of the operating physician, will require a subsequent open or endovascular surgery in the following 30 days.
8. In cases with symptoms of limb-threatening circulatory compromise, ankle-brachial index <0.4, absolute ankle pressure <50 mmHg or absolute toe pressure <30 mmHg.
9. Pulmonary embolism (PE) defined as either massive (systolic blood pressure < 90 mmHg and/or patient on IV vasoactive medication to support blood pressure), or intermediate high-risk PE, as defined by the European Society Guideline on management of PE. Low-risk PE and/or intermediate low-risk PE can be enrolled.
10. Inability to tolerate contemporary venous intervention procedure due to severe dyspnea or acute systemic illness.
11. Allergy or hypersensitivity to any drugs planned for use in the case (including dexamethasone sodium phosphate, iodinated contrast, low molecular-weight heparin, or recombinant tissue plasminogen activator, rtPA, if planned), except for mild-moderate contrast allergies for which steroid pre-medication can be used.
12. History of, or active heparin-induced thrombocytopenia (HIT).
13. Hemoglobin < 8.0 g/dl.
14. INR > 1.6 before starting anticoagulation.
15. Platelets < 100,000/ml.
16. Severe renal impairment (estimated glomerular filtration rate < 30 ml/min).
17. Active bleeding, recent (< 1 mo) GI bleeding, severe liver dysfunction, bleeding diathesis.
18. Recent (< 3 mo) internal eye surgery or hemorrhagic retinopathy.
19. Recent (< 10 days) major surgery, trauma, cardiopulmonary resuscitation, or other invasive procedure which, in the Investigator's discretion, could impair follow-up or study outcomes.
20. Obstetrical delivery <72 hours prior to procedure.
21. Hemorrhagic stroke within the last 365 days.
22. Intracranial/intraspinal bleed within the last 365 days.
23. Intracranial/intraspinal tumor within the last 365 days.
24. Intracranial/intraspinal vascular malformation within the last 365 days.
25. Intracranial/intraspinal aneurysm within the last 365 days.
26. Active symptomatic COVID-19 infection that, in the Investigator's discretion, could impair follow-up or study outcomes.
27. Severe hypertension on repeated readings (systolic blood pressure > 180 mmHg or diastolic blood pressure > 105 mmHg). This can be treated, and blood pressure must be stable before venous access is obtained (systolic blood pressure <140 mmHg).
28. Pregnant or breastfeeding.
29. Life expectancy < 2 years (e.g. due to active cancer).
30. Major thrombus of the inferior vena cava (IVC) (occlusive or near-occlusive) extending at least one centimeter above the common iliac confluence.
31. Inability to obtain venous access.
32. Inability to recanalize the target vein segment with less than 30% residual obstruction due to thrombus.
33. History of ipsilateral venous stent.
34. DVT target length intended for drug treatment exceeds 50 cm.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically relevant primary patency | 6 months
  Rate of freedom from loss of patency (defined as 100% occlusion of unstented vein or 50% stenosis of stented vein measured by duplex ultrasound or angiogram) with associated symptoms
Limit the progression to PTS | 6 months
  PTS rate by Villalta score ≥5.
Rate of freedom from major adverse event (MAE) | 30 days
  Rate of freedom from composite of all-cause death, clinically significant pulmonary embolism, major bleeding, target vessel thrombosis, infection of treatment or insertion site, or AV fistula of treatment site

CONTACTS AND LOCATIONS:
Locations (17):
- United States (15):
  - Providence St. Joseph Hospital, Orange, California
  - Vascular Care Connecticut, Darien, Connecticut
  - HCA Florida JFK Hospital, Atlantis, Florida
  - Baptist Health, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - CIS Clinical Research, Houma, Louisiana
  - Medstar Health Research Institute, Hyattsville, Maryland
  - Englewood Health, Englewood, New Jersey
  - Stony Brook University Hospital, Stony Brook, New York
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - OhioHealth Research Institute, Columbus, Ohio
  - St John Health System, Bartlesville, Oklahoma
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Galway University Hospital, Galway, Ireland
- Guy's and St. Thomas Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No